CLINICAL TRIAL: NCT02586844
Title: Prospective Comprehensive Molecular Profiling In Neuroendocrine Tumors
Acronym: NET-SEQ
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: NET-SEQ
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Neuroendocrine Tumors; Pancreatic Neuroendocrine Tumors
Keywords: NET; PanNET; Molecular profiling; Transcriptome sequencing
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, 3 tubes of whole blood, archival tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neuroendocrine tumors (NETs): Eligible consenting patients will undergo one-time biopsy, during which at least 3 tumors' core samples (total length of at least 6 cm) will be collected. Core tumor biopsies and 3 vials of whole blood and archived tumor specimens will be obtained for genomic testing analysis.
- panNETs: Eligible consenting patients will undergo one-time biopsy, during which at least 3 tumors' core samples (total length of at least 6 cm) will be collected. Core tumor biopsies and 3 vials of whole blood and archived tumor specimens will be obtained for genomic testing analysis.

SUMMARY:
Prospective study to obtain fresh tumor biopsies and three blood samples from patients with a confirmed histological or cytological diagnosis of well-differentiated neuroendocrine tumors (NETs) or well-differentiated pancreatic neuroendocrine tumors (PanNETs) for molecular profiling.

DETAILED DESCRIPTION:
In this prospective study the aim is to obtain fresh tumor biopsies and three blood samples from patients with a confirmed histological or cytological diagnosis of well-differentiated neuroendocrine tumors (NETs) or well-differentiated pancreatic neuroendocrine tumors (PanNETs). Eligible population includes: NETs and PanNETs patients who have undergone or are undergoing treatment with targeted therapies and have shown prolonged clinical benefit, and NETs and PanNETs patients who have been treated with these agents and just recently progressed. RNA and DNA from fresh tumor biopsies and from mononuclear blood cells will be subjected to transcriptome sequencing and DNA sequencing analyses to evaluate possible genes of interest and related targetable pathways. Moreover, archived tumor samples will be requested from all patients to perform additional genomic testing. Remaining RNA and DNA will be banked for additional exploratory analyses (e.g. further genomic testing, or DNA copy number analysis, or epigenetic evaluations).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Histological or cytological proof of NETs or PanNETs.
* At least one biopsiable lesion deemed medically accessible and safe to biopsy.
* Current/recent treatment with targeted therapies with confirmed clinical benefit; confirmed progression disease to targeted therapies at the time of study enrollment.
* Fulfills local institution's laboratory parameters for tumor biopsy.
* Willingness and ability of patient to provide signed voluntary informed consent.

Exclusion Criteria:

* Any condition that could interfere with their ability to provide informed consent such as dementia or severe cognitive impairment.
* Any contraindication to undergoing a biopsy or blood collection procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histological or cytological diagnosis of NET and PanNET; have at least one biopsiable lesion deemed medically accessible and safe to biopsy; fulfill local institution's laboratory parameters for tumor biopsy, and provided written voluntary informed consent.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
To prospectively collect tumor tissue and blood sample from patients with carcinoid tumors and islet cell tumors. | 3 years

SECONDARY OUTCOMES:
To evaluate gene alterations differences between carcinoid tumors and islet cell tumors. | 3 years
To correlate genomic findings with treatment and clinical outcome. | 3 years
To compare acquired data with existent available databases of whole genome or exome of neuroendocrine tumors | 3 years
To bank remaining samples for additional exploratory analyses (e.g. further genomic testing, or DNA copy number analysis, or epigenetic evaluations). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada